CLINICAL TRIAL: NCT07112222
Title: A Phase I/II, First-in-Human (FIH), Open-Label, Multiple Centre Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetics, Immunogenicity and Preliminary Efficacy of LM-350 in Patients With Advanced Solid Tumors
Brief Title: A Study of LM-350 in Subjects With Advanced Solid Tumours
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: LaNova Medicines Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: LM350-01-101
Record Dates: First submitted 2025-07-16; First posted 2025-08-08 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Malignant Tumors
MeSH Terms: conditions — Neoplasms | interventions — Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Phase I Dose Escalation Part and Dose Confirmation Part (Experimental)
  Interventions: Drug: LM-350 for injection

INTERVENTIONS:
Drug: LM-350 for injection — Q3W,Intravenous Drip

SUMMARY:
For Phase I Dose Escalation Stage, to assess the safety and tolerability of LM-350 in patients with advanced solid tumors,determine the maximum tolerated dose (MTD) or optimal biological dose (OBD), and explore the relationship between the biomarkers and the anti-tumor activity of LM-350.

For Phase II Dose Expansion Stage, to assess the preliminary anti-tumor activity of LM-350 in patients with advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who are willing to participate in the study and sign the informed consent form (ICF) prior to any procedure.
2. Participant must be ≥18 years or the legal age of consent at the time of signing the ICF.
3. Eastern Cooperative Oncology Group (ECOG) performance status of 0-1.
4. Life expectancy ≥ 3 months.
5. Patients with advanced solid tumors confirmed by histopathological diagnosis who have failed standard treatment, are intolerant to standard treatment, or for whom standard treatment is currently unsuitable.
6. Pre-treatment archived tumour tissue (within 3 years) or on-treatment tumour biopsy could be provided for biomarker analysis.
7. Must have at least one measurable lesion according to RECIST v1.1.
8. Adequate organ and bone marrow function as defined by protocol.
9. Subjects who are able to communicate well with investigators and understand and adhere to the requirements of this study.

Exclusion Criteria:

1. Participate in any other clinical trial within 28 days prior to 1st dosing of LM-350.
2. Subjects who have received treatment with the same targeting.
3. History of ≥ Grade 3 late diarrhea during or after previous treatment with a topoisomerase inhibitor.
4. Subjects who have received the following anti-tumor treatments within the specified time periods prior to the first dosing of LM-350.
5. Any adverse event from prior anti-tumour therapy has not yet recovered to ≤ grade 1 of CTCAE v5.0.
6. Subjects with uncontrolled tumour-related pain.
7. Subjects with known central nervous system (CNS) or meningeal metastasis.
8. Subjects who have clinically uncontrollable third-space fluid accumulation.
9. Subjects who experienced grade 3 or higher hypersensitivity to the treatment that contains monoclonal antibody.
10. Subjects who take systemic corticosteroids (≥ 10 mg/day of prednisone or equivalents) or other systemic immunosuppressive medications within 2 weeks prior to the first dose of LM-350.
11. Has a history of (noninfectious) ILD/pneumonitis that required steroids, has current ILD/pneumonitis, or where suspected ILD/pneumonitis cannot be ruled out by imaging at Screening.
12. Clinically severe pulmonary compromise resulting from intercurrent pulmonary illnesses, and any autoimmune, or prior pneumonectomy.
13. Use of any live attenuated vaccines within 28 days prior to 1st dosing of LM-350.
14. Current unstable of full-dose oral or parenteral anticoagulants or thrombolytic agents for > 2 weeks prior to the first dose of LM-350.
15. Subjects with active or a documented history of chronic inflammatory bowel disease (ulcerative colitis, Crohn's disease).
16. Subjects with complete or incomplete intestinal obstruction within 3 months prior to the first dose of the study drug , orpatients who are currently at the risk of intestinal perforation.
17. Subjects who received major surgery or interventional treatment within 28 days prior to 1st dosing of LM-350.
18. Subjects who have severe cardiovascular disease.
19. Subjects who have uncontrolled or severe illness.
20. Subjects who have a history of immunodeficiency disease.
21. HIV infection, active infection including tuberculosis, HBV and HCV infection.
22. Subjects who have other active malignancies which are likely to require the treatment.
23. Child-bearing potential female who have positive results in pregnancy test or are lactating.
24. Subjects who have psychiatric illness or disorders that may preclude study compliance.
25. Subject who is judged as not eligible to participate in this study by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-08-28 (Actual); Primary Completion 2028-06-30 (Estimated); Study Completion 2030-06-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of dose-limitingtoxicity (DLT) | 78 weeks
  Phase I
Incidence of Treatment-Emergent Adverse Events (AEs) | 78 weeks
  Phase I
Incidence of serious adverse events (SAEs) | 78 weeks
  Phase I
Temperature (Celsius) | 78 weeks
  Phase I
Pulse in BPM(Beat per Minute) | 78 weeks
  Phase I
Blood Pressure in mmHg | 78 weeks
  Phase I
Weight in Kg | 78 weeks
  Phase I
Height in centimeter | 78 weeks
  Phase I
Blood Routine examination -> Complete Blood Count | 78 weeks
  Phase I
Urine Routine examination ->Urinalysis | 78 weeks
  Phase I
Blood Biochemistry test -> Electrolytes and Metabolic Parameters | 78 weeks
  Phase I
Coagulation function test-For the detection of Prothrombin time (PT), Activated partial thromboplastin time (APTT), International normalized | 78 weeks
  Phase I
Pregnancy test | 78 weeks
  Phase I
Echocardiography- LVEF(Left Ventricular Ejection Fraction) in percentage | 78 weeks
  Phase I
12-lead electrocardiogram (ECG) in HR | 78 weeks
  Phase I
12-lead electrocardiogram (ECG) in RR | 78 weeks
  Phase I
12-lead electrocardiogram (ECG) in QRS | 78 weeks
  Phase I
12-lead electrocardiogram (ECG) in QT | 78 weeks
  Phase I
12-lead electrocardiogram (ECG) in QTcF | 78 weeks
  Phase I
ECOG(Eastern Cooperative Oncology Group) score | 78 weeks
  Phase I
Objective Response Rate (ORR) | 130 weeks
  Phase II

SECONDARY OUTCOMES:
Pharmacokinetic (PK) Parameter: Maximum Observed Concentration (Cmax) | 130 weeks
  Phase I/II
PK Parameter:Time of Maximum Observed Concentration (Tmax) | 130 weeks
  Phase I/II
PK Parameter: Area Under the Concentration-time Curve(AUC) | 130 weeks
  Phase I/II
PK Parameter: Steady State Maximum Concentration(Cmax,ss) PK Parameter: Steady State Maximum Concentration(Cmax,ss) | 130 weeks
  Phase I/II
PK Parameter: Steady State Minimum Concentration(Cmin,ss) | 130 weeks
  Phase I/II
PK Parameter: Systemic Clearance at Steady State (CLss) | 130 weeks
  Phase I/II
PK Parameter: Accumulation Ratio (Rac) | 130 weeks
  Phase I/II
PK Parameter: Elimination Half-life (t1/2) | 130 weeks
  Phase I/II
PK Parameter: Volume of Distribution at Steady-State (Vss) | 130 weeks
  Phase I/II
PK Parameter: Degree of Fluctuation (DF) | 130 weeks
  Phase I/II
Immunogenicity testing->Anti-Drug Antibody test | 130 weeks
  Phase I/II
Objective Response Rate (ORR) | 130 weeks
  Phase I
Duration of Response (DOR) in Month | 130 weeks
  Phase I/II
Disease control rate (DCR) in percentage | 130 weeks
  Phase I/II
Progression-free survival (PFS) in Month | 130 weeks
  Phase I/II
Overall survival (OS) in Month | 130 weeks
  Phase I/II
Changes of target lesions from baseline in Millimeter | 130 weeks
  Phase I/II
Incidence of adverse events (AEs) | 130 weeks
  Phase II
Incidence of serious adverse events (SAEs) | 130 weeks
  Phase II
Temperature (Celsius) | 130 weeks
  Phase II
Pulse in BPM(Beat per Minute) | 130 weeks
  Phase II
Blood Pressure in mmHg | 130 weeks
  Phase II
Weight in Kg | 130 weeks
  Phase II
Height in centimeter | 130 weeks
  Phase II
Blood Routine examination -> Complete Blood Count | 130 weeks
  Phase II
Urine Routine examination ->Urinalysis | 130 weeks
  Phase II
Blood Biochemistry test -> Electrolytes and Metabolic Parameters | 130 weeks
  Phase II
Coagulation function test-For the detection of Prothrombin time (PT), Activated partial thromboplastin time (APTT), International normalized ratio (INR) | 130 weeks
  Phase II
Pregnancy test | 130 weeks
  Phase II
Echocardiography- LVEF(Left Ventricular Ejection Fraction) in percentage | 130 weeks
  Phase II
ECOG(Eastern Cooperative Oncology Group) score | 130 weeks
  Phase II
12-lead electrocardiogram (ECG) in HR | 130 weeks
  Phase II
12-lead electrocardiogram (ECG) in RR | 130 weeks
  Phase II
12-lead electrocardiogram (ECG) in PR | 130 weeks
  Phase II
12-lead electrocardiogram (ECG) in QRS | 130 weeks
  Phase II
12-lead electrocardiogram (ECG) in QT | 130 weeks
  Phase II
12-lead electrocardiogram (ECG) in QTcF | 130 weeks
  Phase II
Biomarker test -> Tumor tissue biomarker test | 130 weeks
  Phase I/II

CONTACTS AND LOCATIONS:
Locations (4):
- Australia (3):
  - Cancer Care Wollongong Pty Limited, Wollongong, New South Wales
  - Cancer Research SA, Adelaide, South Australia
  - Peninsula and South Eastern Haematology and Oncology Group, Frankston, Victoria
- Beijing Cancer Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No